CLINICAL TRIAL: NCT00972335
Title: A Phase II Trial of the Combination of Bevacizumab and Everolimus in Patients With Refractory, Progressive Intracranial Meningioma
Brief Title: Trial of the Combination of Bevacizumab and Everolimus in Patients With Refractory, Progressive Intracranial Meningioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to slow accrual
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CNS 12
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Intracranial Meningioma
Keywords: Avastin; RAD001; Meningioma; Bevacizumab; Everolimus; Brain
MeSH Terms: conditions — Meningioma | interventions — Everolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): Everolimus; this drug will be dosed at 10 mg orally DAILY for the duration of the study.
  Bevacizumab; this drug will be given IV at 10 mg/kg on Days 1 and 15 of each 28-day treatment cycle for the duration of the study
  Interventions: Drug: Everolimus; Drug: Bevacizumab

INTERVENTIONS:
Drug: Everolimus — This drug will be dosed at 10 mg orally DAILY for the duration of the study.
  Other Names: RAD001
Drug: Bevacizumab — This drug will be given IV at 10 mg/kg on Days 1 and 15 of each 28-day treatment cycle for the duration of the study.
  Other Names: Avastin

SUMMARY:
In this multicenter, Phase II trial, the investigators plan to evaluate the activity of the combination of bevacizumab and everolimus in patients with recurrent, progressive meningioma following maximal treatment with surgical resection and local radiation therapy. Although these patients are relatively rare, there is currently no established standard of treatment for a disease that causes a great deal of morbidity, and that is eventually fatal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age.
2. Histologic diagnosis of meningioma, WHO grade 1, 2, or 3 (benign, atypical, or malignant). In addition, patients with definitive radiologic evidence of meningioma who are unresectable, and in whom radiation therapy without biopsy is the standard treatment, are also eligible.
3. All patients must have developed recurrent disease/progression after receiving all standard treatments, which must include the following:

   * surgical resection, if possible;
   * definitive radiation therapy for unresectable meningioma, or for recurrent meningioma after resection.
   * patients must be at least 4 weeks post-surgery, and must be at least 2 weeks post-radiation therapy, with resolution of related toxicities.
4. All patients must have progressive symptoms judged to be directly related to their recurrent/progressive meningioma. Patients with no new symptoms, or patients with stable neurologic deficits from previous surgical resection, are not eligible.
5. Patients may have had 0 or 1 previous systemic treatment regimens.
6. ECOG performance status of 0-2.
7. Adequate bone marrow, kidney, and liver function, as follows:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥9 g/dL
   * Platelets ≥100,000/L (≤7 days prior to treatment)
   * AST or ALT ≤2.5 x institutional upper limit of normal (ULN)
   * Total bilirubin ≤1.5 x institutional ULN
   * Serum creatinine ≤1.5 x institutional ULN
8. Life expectancy of at least 12 weeks.
9. Ability to swallow whole pills.
10. Patients must have measurable disease on MRI scan.
11. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
12. INR ≤1.5 x institutional upper limit of normal (ULN) . (Anticoagulation is allowed if target INR is ≤1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at the time of study entry).
13. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x institutional ULN. Note: In case one or both of these thresholds are exceeded, the patient can only be included in the study after initiation of appropriate lipid-lowering medication.
14. Patients must be accessible for treatment and follow-up.
15. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Previous treatment with bevacizumab or any other anti-angiogenesis agents.
2. Previous treatment with m-TOR inhibitors (sirolimus, temsirolimus, everolimus).
3. Patients who have had major surgery or significant traumatic injury within 4 weeks of the start of study drugs, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients that may require major surgery during the course of the study.
4. Minor surgical procedures (with the exception of the placement of portacath or other central venous access) must be completed at least 7 days prior to beginning protocol treatment.
5. Women who are pregnant or lactating.
6. Patients with proteinuria at screening as demonstrated by either:

   urine protein creatinine (UPC) ratio 1.0 at screening OR urine dipstick for proteinuria 2+ (patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection, and must demonstrate 1 g of protein/24 hours to be eligible)
7. Patients with a serious non-healing wound, active ulcer, or untreated bone fracture.
8. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
9. Patients with history of hematemesis or hemoptysis (defined as having bright red blood of ½ teaspoon or more per episode) within 1 month prior to study enrollment.
10. History of myocardial infarction or unstable angina within 6 months of beginning treatment.
11. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and /or diastolic blood pressure >100 mmHg while on antihypertensive medications).
12. New York Heart Association (NYHA) class II or greater congestive heart failure (CHF).
13. Serious cardiac arrhythmia requiring medication.
14. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of treatment.
15. History of stroke or transient ischemic attack within 6 months prior to beginning treatment.
16. Any prior history of hypertensive crisis or hypertensive encephalopathy.
17. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1 of beginning treatment.
18. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
19. Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

    * unstable angina pectoris, symptomatic CHF, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
    * severely impaired lung function
    * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
    * active (acute or chronic) or uncontrolled severe infections
    * liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
20. Known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus), or to its excipients.
21. Immunization with attenuated live vaccines within 1 week of the study, or anytime during study treatment.
22. Chronic, systemic treatment with immunosuppressive agents. Patients who require a stable dose of corticosteroids for control of cerebral edema are eligible. Topical or inhaled steroids are also allowed.
23. Known human immunodeficiency virus (HIV) infection.
24. Grapefruits, star fruits, seville oranges, and their juices and products, should be avoided.
25. Drugs or substances known to be inhibitors or inducers of the isoenzyme CYP3A4 should be avoided.
26. Use of St. John's Wort or rifampicin.
27. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
28. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
29. Use of any non-approved or investigational agent within 4 weeks of study entry. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
30. Other malignancies within the last 3 years, with the exception of adequately treated basal or squamous cell carcinomas of the skin, or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Florida Hospital Cancer Insitute, Orlando, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Cancer Insititute Memphis, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 17 (One patient was enrolled but showed no evidence of disease at study entry and was not treated)
Completed | 0 (Patients were on study until an event or condition occured which required them to come off study)
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: All treated patients (one enrolled patient was not treated)
Arm/Group | Combination Therapy
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS), in the Treatment of Patients With Refractory Meningioma.
Description: Progression-free survival (PFS) is defined as the time from randomization until objective tumor progression (PD) or death. Progression is defined per MacDonald criteria for response as ≥25% increase in size of enhancing tumor or any new tumor on MRI scan, neurologically worse, and steroids stable or increased.
Time Frame: 18 months
Population: Includes all enrolled and treated patients (one patient not treated)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 17
months | 22 [4.5 to 26.8]

2. Secondary Outcome: To Evaluate the Toxicity of Bevacizumab/Everolimus in Patients With Recurrent Meningioma.
Time Frame: 18 months
Population: Includes all treated patients (one patient not treated)
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 17
participants
  Thrombocytopenia | 9
  Anemia | 6
  Leukopenia | 2
  Neutropenia | 2
  Hypercholesterolemia | 9
  Mucositis | 9
  Fatigue | 8
  Proteinuria | 6
  Hypertriglyceridemia | 6
  Rash/desquamation | 6
  Diarrhea | 6
  Hypertension | 5
  Edema-limb | 5
  Vomiting | 4
  Anorexia | 4
  Nausea | 4
  Hyperglycemia | 3
  Pain - oral cavity | 3
  Epistaxis | 3
  Headache | 3
  Arthralgia | 3

3. Secondary Outcome: To Correlate the Activity of This Treatment Regimen With Expression of Selected Intra-tumoral Biomarkers.
Time Frame: 18 months
Population: The results were not analyzed at study closure as the data were not collected.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=17)
Ataxia (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
General disorders and administration site conditions - Other, disease progression (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Infections and infestations - Other, pneumonia (Infections and infestations) | 1
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 2
Seizure (Nervous system disorders) | 1
urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=17)
Fatigue (General disorders) | 12
Headache (Nervous system disorders) | 11
Mucositis (Gastrointestinal disorders) | 10
Platelet count decreased (Investigations) | 10
Cholesterol high (Investigations) | 9
Anemia (Blood and lymphatic system disorders) | 8
Diarrhea (Gastrointestinal disorders) | 8
Proteinuria (Renal and urinary disorders) | 8
Hypertension (Vascular disorders) | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Edema limbs (General disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5
Memory impairment (Nervous system disorders) | 5
Alanine aminotransferase increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Insomnia (Psychiatric disorders) | 4
Neutrophil count decreased (Investigations) | 4
Infections and infestations - Other, pneumonia (Infections and infestations) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Depression (Psychiatric disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 3
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
neck pain (Musculoskeletal and connective tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 2
Upper respiratory infection (Infections and infestations) | 2
Seizure (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Creatinine increased (Investigations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema (General disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Eye disorders - Other, vision changes (Eye disorders) | 1
Flu like symptoms (General disorders) | 1
Gastrointestinal disorders - Other, stomatitis (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, disease progression (General disorders) | 1
Heart Failure (Cardiac disorders) | 1
Hematoma (Vascular disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nervous system disorders - Other, speech impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Renal and urinary disorders - Other, renal failure (Renal and urinary disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Wound complication (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Enrollment closed early due to slow accrual, leading to small number of subjects analyzed - biomarker analysis outcome measure not analyzed or reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites